CLINICAL TRIAL: NCT06253442
Title: A Comparative Study Between Ultrasound Guided Interscalene Block and Combined Ultrasound Guided Suprascapular and Axillary Nerve Blocks for Proximal Humerus Fracture Surgeries.
Brief Title: Comparison Between Interscalene Block and Combined Suprascapular and Axillary Blocks for Proximal Humerus Fracture Surgeries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, riham fathy galal, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAMSU R10/2024
Record Dates: First submitted 2024-01-30; First posted 2024-02-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Proximal Humerus Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients will receive Supra scapular nerve block and Axillary nerve block. (Active Comparator): ultrasound guided suprascapular nerve block combined with ultrasound guided axillary nerve block will be provided to the patient
  Interventions: Procedure: Patients will receive Supra scapular nerve block and Axillary nerve block.
- Patients will receive Interscalene block. (Active Comparator): ultrasound guided interscalene brachial plexus block will be provided to the patient
  Interventions: Procedure: Patients will receive Interscalene block.

INTERVENTIONS:
Procedure: Patients will receive Supra scapular nerve block and Axillary nerve block. — Suprascapular nerve block will be done by posterior approach with the patient sitting up and leaning forward. The linear ultrasound probe will identify the suprascapular nerve, after that we will inject aliquots of Sunnypivacaine 0.5% 15 ml after negative aspiration of blood.
  For the axillary nerve block, the ultrasound transducer will be placed in a sagittal plane over the humeral head on the posterior aspect of the arm to identify the deltoid muscle, neck of the humerus, the teres minor muscle, the circumflex humeral artery, and the triceps muscle. After the neurovascular quadrangular space identification and observing the deltoid muscle response to stimulation, a local anesthetic (10 ml 0.25% Sunnypivacaine) will be injected with the in-plain technique.
  Arms: Patients will receive Supra scapular nerve block and Axillary nerve block.
Procedure: Patients will receive Interscalene block. — Interscalene nerve block will be done ultrasound-guided using a linear array ultrasound transducer. While the patient is in the supine position, the head will be rotated to the contralateral side of the block. Ultrasound scanning will be performed in the transverse plane with long axis of the probe parallel to clavicle to visualize the brachial plexus between the anterior and middle scalene muscles. A 5-cm 22-gauge insulated needle will then be inserted in line with the probe in a lateral-to-medial needle orientation. Local anesthetic solution will then be injected in 15-ml aliquots Sunnypivacaine 0.5% after negative aspiration for blood to achieve spread posterior to or between the C5 and C6 nerve roots.
  Arms: Patients will receive Interscalene block.

SUMMARY:
A Comparative study Between Ultrasound guided Interscalene Block and Combined Ultrasound guided suprascapular and axillary nerve blocks for proximal humerus fracture Surgeries.

The aim of this study is to investigate whether (Suprascapular nerve block) and (Axillary nerve block) are effective in providing analgesia for shoulder surgery as an (Interscalene block), while minimizing the occurrence of hemi-diaphragmatic paralysis. We hypothesized that analgesia with a (Suprascapular nerve block and Axillary nerve block) would be noninferior compared with patients receiving an interscalene block and the incidence of hemi-diaphragmatic paralysis would be significantly lower with (Suprascapular nerve block and Axillary nerve block) in proximal humerus fracture surgeries.

DETAILED DESCRIPTION:
A Comparative study Between Ultrasound guided Interscalene Block and Combined Ultrasound guided suprascapular and axillary nerve blocks for proximal humerus fracture Surgeries.

The aim of this study is to investigate whether (Suprascapular nerve block) and (Axillary nerve block) are effective in providing analgesia for shoulder surgery as an (Interscalene block), while minimizing the occurrence of hemi-diaphragmatic paralysis. We hypothesized that analgesia with a (Suprascapular nerve block and Axillary nerve block) would be noninferior compared with patients receiving an interscalene block and the incidence of hemi-diaphragmatic paralysis would be significantly lower with (Suprascapular nerve block and Axillary nerve block) in proximal humerus fracture surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Patients American Society of anesthesiologists' physical status (ASA) I to II.
2. Aged 18 to 65 years.
3. Both sexes.
4. Patients scheduled for proximal humerus fracture surgeries.

Exclusion Criteria:

1. Patient refusal
2. ASA physical status III or more.
3. Patients with known allergy to any of the study drugs.
4. Infection at the site of injection.
5. Patients with history of cardiovascular disease.
6. Patients with renal disease.
7. Patients with hepatic disease.
8. Patients with neuromuscular disease.
9. Presence of any coagulopathy.
10. Chronic opioid, gabapentin or pregabalin use.
11. Patients with history of any psychiatric disorder.
12. BMI more than 35 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Individual visual analog pain scores (VAS) at 0, 6, 12 and 24 h postoperatively (VAS; 0 = no pain and 10 = worst pain imaginable). | 24 HOURS
  Individual visual analog pain scores (VAS) at 0, 6, 12 and 24 h postoperatively (VAS; 0 = no pain and 10 = worst pain imaginable).
The presence of moderate-to-severe pain, defined as visual analog pain scores (VAS) 4 or greater during the first 24 h postoperative. | 24 HOURS
  The presence of moderate-to-severe pain, defined as visual analog pain scores (VAS) 4 or greater during the first 24 h postoperative.
Time to first reported pain and first analgesic request during post-anesthesia care unit stay (in minutes). | 24 HOURS
  Time to first reported pain and first analgesic request during post-anesthesia care unit stay (in minutes).
Analgesic consumption during surgery, in post-anesthesia care unit, and during the first 24 h post-surgery. | 24 hours
  Analgesic consumption during surgery, in post-anesthesia care unit, and during the first 24 h post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No